CLINICAL TRIAL: NCT07404787
Title: SAFEGUARD Phase 2 Pathfinding Study
Brief Title: Evaluation of a Telehealth Case Management Intervention to Prevent Suicide Among Soldiers Discharged From Psychiatric Hospitalization
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Uniformed Services University of the Health Sciences (U.S. Federal Agency)
Collaborators: Harvard Medical School (HMS and HSDM) (Other); University of Michigan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: USUHS.2025-156; Federal Award # HU00012520025 (Other Grant/Funding Number: Office of the Assistant Secretary of Defense for Health Affairs)
Record Dates: First submitted 2026-02-04; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-01

CONDITIONS: Suicide; Suicide Attempt
Keywords: suicide; suicide attempt; hospital discharge; military; intervention; case management
MeSH Terms: conditions — Suicide; Suicide, Attempted | interventions — Axon Guidance; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pathfinding intervention plus Treatment As Usual (TAU) (Experimental): Pathfinding is a 6-month, adjunctive, telehealth intervention that integrates 2 evidence-based case management programs and adapts them for active duty soldiers: Coping Long Term with Active Suicide Program (CLASP), a case management intervention for suicidal patients transitioning out of psychiatric hospitals; and Critical Time Intervention (CTI), a more general case management intervention for high-risk transitions out restrictive environments. Administered remotely by a centrally trained & supervised team of "Guides." Focuses on key suicide risk factors (e.g., treatment engagement, social connection, problem-solving) and unmet needs across life domains (e.g., legal, financial, housing, and relationships). Participants receive Pathfinding in addition to standard post-discharge care (see TAU intervention description for details).
  Interventions: Behavioral: Pathfinding
- Treatment As Usual (TAU) (Active Comparator): Treatment As Usual (TAU) is the Army's standard care for soldiers discharged from inpatient psychiatric treatment. It involves discharge planning, risk assessment, and referrals (as detailed in the TAU intervention description).
  Interventions: Behavioral: Treatment As Usual (TAU)

INTERVENTIONS:
Behavioral: Pathfinding — The Pathfinding intervention consists of remote (videoconference or phone) interactions between participants and masters-level Guides over the 6 months following study enrollment. Participants have the option of involving a support person (SP) in the intervention (e.g., family member, friend). First 4 sessions (45 min. each) occur as soon as possible following hospital discharge and focus on orientation to Pathfinding, identifying a SP, and identifying and prioritizing values/needs, values-consistent goals, corresponding actions, and relevant resources. Participants subsequently receive up to 10 brief (15-30 min. each) contacts to monitor risk and progress. Frequency of contacts is front-loaded and diminishes over time as participants take more control over managing their transition. SPs are contacted for up to 5 sessions (10-15 min. each) to help with monitoring and support. Sessions, risk assessments, and any crisis response actions are documented in the electronic health record.
  Arms: Pathfinding intervention plus Treatment As Usual (TAU)
Behavioral: Treatment As Usual (TAU) — TAU is standard post-discharge care based on Defense Health Agency policy (DHA Administrative Instruction 6025.06): Discharge plans must consist of referral with plans for outpatient or partial hospitalization follow-up within 7 days (optimally within 72 hours). Discharged patients are placed on a High-Risk (HR) list for at least 30 days. During this period, patients are seen weekly for follow-up appointments or attendance of the HR group if individual psychotherapy is not available. If, after 4 weeks, the patient is assessed as no longer acutely suicidal, they are removed from the HR list. After removal from the HR list, patients are seen either weekly or every other week, depending on clinical need. Initial care coordination is handled by the discharge nurse. Ongoing care coordination is managed by the outpatient mental health team. Safety planning is conducted at discharge and every few sessions thereafter using the DHA safety plan. Safety assessments are conducted at each visit.
  Arms: Treatment As Usual (TAU)

SUMMARY:
This study evaluates the effectiveness of Pathfinding, a 6-month, remotely-delivered case management intervention designed to decrease suicidal behavior among active-duty Regular Army soldiers recently discharged from inpatient psychiatric treatment. Soldiers discharged from military treatment facilities across the U.S. will be identified and recruited to participate. Those who consent will be randomly assigned to receive either Treatment As Usual (TAU), which is the Army's standard post-discharge care, or TAU plus Pathfinding. Participants will complete a baseline assessment and follow-up assessments 6 months and 12 months later. The 6- and 12-month follow-up periods will also include examination of participants' electronic healthcare data and Army administrative data. The overall goals of the study are: (1) to evaluate whether Pathfinding decreases suicidal behaviors among soldiers transitioning from psychiatric hospitalization back to the community; and (2) to determine which discharged soldiers are most likely to benefit from the Pathfinding intervention versus TAU alone.

DETAILED DESCRIPTION:
Discharge from psychiatric hospitalization is the highest risk period for death by suicide. Intensive case management programs have been effective in reducing post-discharge suicidal behavior, but such programs are too resource-intensive to implement for all psychiatric inpatients. It would be more scalable to target the intervention to those most likely to benefit and implement it remotely with centralized training & management. This study evaluates the effectiveness of Pathfinding, a 6-month, adjunctive, telehealth case management intervention, in decreasing suicide-related behaviors among active-duty Regular Army soldiers over the 12 months following discharge from inpatient psychiatric treatment. The Pathfinding intervention combines elements from two case management programs that have been found to reduce suicidal behavior and other negative outcomes among individuals transitioning out of the hospital and back to the community-Coping with Long-Term Active Suicide Program (CLASP) and Critical Time Intervention (CTI)-and adapts them for the unique needs of an active-duty military population. The intervention is delivered remotely by "Guides," masters-level mental health professionals who are centrally trained and supervised.

Soldiers hospitalized for inpatient psychiatric care at military treatment facilities (MTFs) across the U.S. will be identified in the electronic health record (EHR) as soon as possible after being discharged. A previously developed machine learning model based on EHR and Army administrative data will be used to stratify discharged soldiers based on their predicted probability of suicidal behavior. Soldiers will be recruited from across the distribution of predicted risk via emails, text messages, and phone calls. Consenting soldiers will complete a baseline assessment of their health, experiences, and characteristics. They will then be randomized to receive either Treatment As Usual (TAU), which is the Army's standard post-discharge care, or TAU plus the 6-month Pathfinding case management intervention. All participants will be administered follow-up assessments 6 and 12 months after baseline to identify self-reported suicide-related events and other outcomes. Outcomes will also be tracked through EHR data.

The study will examine: (1) whether Pathfinding decreases suicide-related behaviors among soldiers transitioning from psychiatric hospitalization back to the community; and (2) whether certain soldiers are more likely than others to benefit from the Pathfinding intervention versus TAU alone.

ELIGIBILITY:
Inclusion Criteria:

* Active duty Regular Army soldiers recently discharged from inpatient psychiatric care at a military treatment facility in the US
* Access to telephone and computer (including smartphone)

Exclusion Criteria:

* Impaired ability to provide informed consent
* Terminal illness
* Failure to complete baseline survey within 30 days of discharge
* Positive screen for post-discharge suicide-related behaviors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2026-02-11 (Estimated); Primary Completion 2028-08-31 (Estimated); Study Completion 2029-08-31 (Estimated)

PRIMARY OUTCOMES:
Suicide-related behaviors | Within the 12 months following completion of the baseline assessment
  Suicide-related behaviors are defined as: suicide death (administratively documented or informant reported), nonfatal suicide attempt (self-reported or administratively documented), and interrupted suicide attempt, aborted suicide attempt, and preparatory behaviors for suicide (the latter 3 are all self-reported).

SECONDARY OUTCOMES:
Number of suicide attempts | Within the 12 months following completion of the baseline assessment
  A count of nonfatal suicide attempts (self-reported or administratively documented) that occurred during the follow-up period.
Rehospitalization | Within the 12 months following completion of the baseline assessment
  Psychiatric hospitalization (self-reported, informant reported, or administratively documented) during the follow-up period.
Non-suicide death | Within the 12 months following completion of the baseline assessment
  Any manner of death other than suicide (informant reported or administratively documented) during the follow-up period.
Risky behaviors | Within the 12 months following completion of the baseline assessment
  Risky behaviors (self-reported) related to driving or riding in a vehicle, sexual encounters, and aggression (bullying, sexual harassment, intimate partner violence) during the follow-up period.
Suicide ideation | Within the 12 months following completion of the baseline assessment
  Worst-week frequency, severity, and controllability of suicide ideation during the follow-up period.
Low psychological resilience | Within the 12 months following completion of the baseline assessment
  Perceived increase or decrease in ability to manage stressful experiences (self-reported) during the follow-up period.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Herman, D. B., Susser, E. S., & Conover, S. (2024). Critical Time Intervention: Mobilizing Supports for People During Perilous Transitions. Oxford University Press.
- [Background] Miller, I., Gaudiano, B., & Weinstock, L. (2022). The Coping Long Term with Active Suicide Program (CLASP): A multi-modal intervention for suicide prevention. Oxford University Press.
- [Background] Miller IW, Gaudiano BA, Weinstock LM. The Coping Long Term with Active Suicide Program: Description and Pilot Data. Suicide Life Threat Behav. 2016 Dec;46(6):752-761. doi: 10.1111/sltb.12247. Epub 2016 Apr 2. PMID 27038050
- [Background] Weinstock LM, Bishop TM, Bauer MS, Benware J, Bossarte RM, Bradley J, Dobscha SK, Gibbs J, Gildea SM, Graves H, Haas G, House S, Kennedy CJ, Landes SJ, Liu H, Luedtke A, Marx BP, Miller A, Nock MK, Owen RR, Pigeon WR, Sampson NA, Santiago-Colon A, Shivakumar G, Urosevic S, Kessler RC. Design of a multicenter randomized controlled trial of a post-discharge suicide prevention intervention for high-risk psychiatric inpatients: The Veterans Coordinated Community Care Study. Int J Methods Psychiatr Res. 2024 Dec;33(4):e70003. doi: 10.1002/mpr.70003. PMID 39352173
- [Background] Kessler RC, Warner CH, Ivany C, Petukhova MV, Rose S, Bromet EJ, Brown M 3rd, Cai T, Colpe LJ, Cox KL, Fullerton CS, Gilman SE, Gruber MJ, Heeringa SG, Lewandowski-Romps L, Li J, Millikan-Bell AM, Naifeh JA, Nock MK, Rosellini AJ, Sampson NA, Schoenbaum M, Stein MB, Wessely S, Zaslavsky AM, Ursano RJ; Army STARRS Collaborators. Predicting suicides after psychiatric hospitalization in US Army soldiers: the Army Study To Assess Risk and rEsilience in Servicemembers (Army STARRS). JAMA Psychiatry. 2015 Jan;72(1):49-57. doi: 10.1001/jamapsychiatry.2014.1754. PMID 25390793
- [Background] Kessler RC, Bauer MS, Bishop TM, Bossarte RM, Castro VM, Demler OV, Gildea SM, Goulet JL, King AJ, Kennedy CJ, Landes SJ, Liu H, Luedtke A, Mair P, Marx BP, Nock MK, Petukhova MV, Pigeon WR, Sampson NA, Smoller JW, Miller A, Haas G, Benware J, Bradley J, Owen RR, House S, Urosevic S, Weinstock LM. Evaluation of a Model to Target High-risk Psychiatric Inpatients for an Intensive Postdischarge Suicide Prevention Intervention. JAMA Psychiatry. 2023 Mar 1;80(3):230-240. doi: 10.1001/jamapsychiatry.2022.4634. PMID 36652267